CLINICAL TRIAL: NCT05987852
Title: Hyperbaric Oxygen Therapy for Ulcerative Colitis Patients Hospitalized for Moderate to Severe Flares: A Multi-Center, Randomized, Double-Blind, Sham-Controlled Trial
Brief Title: Hyperbaric Oxygen Therapy for Ulcerative Colitis (HBOT-UC)
Acronym: HBOT-UC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Lauren C Balmert, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HBOT-UC; 1U01DK134321 (NIH)
Record Dates: First submitted 2023-08-01; First posted 2023-08-14 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis
Keywords: hyperbaric oxygen therapy; HBOT; ulcerative colitis; hyperbaric oxygen
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: 5-day intervention period; 12 months observational period through standard of care visits and follow-up
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Hyperbaric Oxygen Therapy (Experimental): Participants enrolled in the active intervention group receiving HBOT will undergo compression to 2.4 Atmospheres Absolute (ATA; 100% O2) for 90 minutes with two 5-10 minute "air breaks" (breathing room air at the 2.4 ATA) during the session. This is done once a day for 5 days.
  Interventions: Device: Hyperbaric Oxygen Therapy
- Sham Hyperbaric Air (Sham Comparator): This control arm will undergo compression to 1.34 ATA for monoplace chambers and 2.4 ATA for multiplace chambers for the full 90-minute session but 21% oxygen instead of 100% oxygen being administered. These participants will also have two 5-10 minute "air breaks" to mimic the treatment protocol. Multiplace sham sessions will have modified air breaks to avoid decompression sickness. This will happen once a day for 5 days.
  Interventions: Other: Sham Hyperbaric Air

INTERVENTIONS:
Device: Hyperbaric Oxygen Therapy — Participants enrolled in the active intervention group receiving HBOT will undergo compression to 2.4 Atmospheres Absolute (ATA; 100% O2) for 90 minutes with two 5-10 minute "air breaks" (breathing room air at the 2.4 ATA) during the session. This is done once a day for 5 days.
  Arms: Hyperbaric Oxygen Therapy
Other: Sham Hyperbaric Air — This control arm will undergo compression to 1.34 ATA for monoplace chambers and 2.4 ATA for multiplace chambers for the full 90-minute session but 21% oxygen instead of 100% oxygen being administered. These participants will also have two 5-10 minute "air breaks" to mimic the treatment protocol. Multiplace sham sessions will have modified air breaks to avoid decompression sickness. This will happen once a day for 5 days.
  Arms: Sham Hyperbaric Air

SUMMARY:
Chronic intestinal hypoxia and accompanying mucosal inflammation is a hallmark of ulcerative colitis (UC). Hyperbaric oxygen therapy (HBOT) involves breathing 100% oxygen under increased atmospheric pressure to increase tissue oxygenation. Two small prospective randomized controlled trials have demonstrated that the delivery of HBOT to UC patients hospitalized for acute moderate to severe flares results in improved remission rates and avoidance of in-hospital progression to biologics, small molecules, or colectomy. In this larger trial the study aims to confirm the treatment benefits of HBOT for hospitalized UC patients and study the immune-microbe mechanisms underpinning treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Participants with known or newly diagnosed UC who require hospitalization for an acute moderate to severe flare
* Age 18-85
* Able to fully participate in all aspects of the trial
* Consented and able to receive first HBOT session within first 48 hours of initiation of intravenous steroids
* Agreement to not participate in another trial for the duration of the active intervention period

Exclusion Criteria:

* Received hyperbaric oxygen therapy either as part of standard of care or through a clinical trial prior to enrollment
* Complication requiring urgent surgical intervention
* Requirement for new start of a biologic or small molecule during the hospitalization prior to randomization and/or anticipated requirement for rescue medical or surgical therapy within 48 hours of randomization
* Toxic megacolon
* Inability to receive intravenous steroids
* Historically failed or been exposed to 4 or more classes of advanced therapeutic options
* Known or suspected diagnosis of Crohn's colitis, indeterminate colitis, ischemic colitis, radiation colitis, diverticular disease associated with colitis, microscopic colitis or infectious colitis
* Received any investigational drug within 30 days
* Clinically significant cardiac, renal, neurological, endocrine, respiratory or hepatic impairment that increases the risk for HBOT toxicity
* Women who are pregnant or nursing
* Unwillingness to complete course of HBOT

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinical response defined as complete resolution of rectal bleeding and improvement in stool frequency, without need for in-hospital biologics, small molecules, or colectomy by study day 5 | Day 5
  Proportion of participants achieving clinical response as measured by complete resolution of rectal bleeding (Mayo rectal bleeding sub-score of 0) and improvement in stool frequency (at least 1 point reduction in Mayo stool frequency sub-score), without the need for in-hospital biologics, small molecules, or colectomy, by study day 5.

SECONDARY OUTCOMES:
Clinical Response | Day 3
  Sum of Mayo rectal bleeding and stool frequency sub-scores (Key secondary endpoint)
Change in inflammation, as measured by C-reactive protein | Day 3
  Change in inflammation, as measured by C-reactive protein (Key secondary endpoint)
Endoscopic response | Day 5
  Ulcerative Colitis Endoscopic Index of Severity (UCEIS) (Key secondary endpoint)
Steroid-free, colectomy-free, clinical remission | Day 90
  Proportion of participants steroid-free, colectomy-free, and with clinical remission (Full Mayo ≤ 2, with no sub-score > 1)
Endoscopic Improvement | Day 90
  Proportion of participants achieving endoscopic improvement (Mayo endoscopic sub-score of 0 or 1)
Endoscopic Remission | Day 90
  Proportion of participants achieving Endoscopic remission (Mayo endoscopic sub-score of 0)
Mucosal Healing | Day 90
  Proportion of participants achieving Mucosal Healing (Endoscopic sub-score 0 or 1 + Geboes histology score ≤ 2)
Clinical Remission | Day 5
  Proportion of participants achieving clinical remission (Full Mayo ≤ 2, with no sub-score > 1)
Colectomy | Day 90; 12 month
  Proportion of participants requiring colectomy
Re-hospitalization for ulcerative colitis flare | 12 months
  Proportion of participants with re-hospitalization during the follow-up period for ulcerative colitis flare
Numeric Urgency Rating Score | Day 3
  Score ranges from 0-10 ; higher scores are worse
Serious Infections or Serious Adverse Events | Day 5
  Proportion of participants experiencing any serious infections or serious adverse events during intervention period

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Balmert Bonner, PhD, Principal Investigator — Northwestern University
Locations (13):
- United States (13):
  - University of Alabama Medicine, Birmingham, Alabama
  - University of Los Angeles Health, Los Angeles, California
  - University of Miami Health, Miami, Florida
  - Orlando Health, Orlando, Florida
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - University of Louisville, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cornell University Medical Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Allegheny Health, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Dataset with National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Repository.
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Derived] Bonner LB, Sadler C, Lindholm P, Scholtens DM, Dulai PS; HBOT-UC Consortium. Hyperbaric oxygen therapy for ulcerative colitis patients hospitalized for moderate to severe flares (HBOT-UC): study protocol for a multi-center, randomized, double-blind, sham-controlled trial. Trials. 2025 Jun 22;26(1):220. doi: 10.1186/s13063-025-08932-5. PMID 40545548